Н

## CLINICAL STUDY PROTOCOL

STEREOTACTIC BODY RADIOTHERAPY (SBRT) FOR THE TREATMENT OF Protocol Title: A PROSPECTIVE TRIAL OF IMMUNOTHERAPY AND METASTATIC LUNG CANCER: SBRT SENSITIZATION OF THE PROGRAMMED DEATH-I (PD-I) EFFECT

VERSION 6.0, 06/18/2018

Clinical Phase: Pilot/Phase II

Increased response should translate to increased progression free survival and improved Hypothesis: The addition of Stereotactic Body Radiation Therapy sequenced prior to PD-I/PDLI blockade leads to increased immunogenicity and immune system response. survival relative to PD-I blockade monotherapy in metastatic lung cancer.

Principal Investigator

Rachelle M. Lanciano MD

Department of Radiation Oncology

Crozer Keystone Health System/Philadelphia CyberKnife Center

2010 West Chester Pike, Havettown, PA 19083

Confidential: This document contains confidential information that is the property of Precision Radiation Oncology and must not be disclosed to anyone other than designees of Precision Radiation Oncology for conduct of the study, clinical investigators and members of the Institutional Review Board.

#### 1. INTRODUCTION

highly effective and complementary approach to the therapeutic mainstays of surgery, cytotoxic Enhancement of the anti-tumor immune response with immunotherapy agents has emerged as a responses and dramatic tumor regression suggests that immunotherapy may convert previously chemotherapy, targeted drugs and radiation therapy. More recently, the induction of lasting fatal diseases into chronic manageable situations.

hallmark feature of cancer progression and carcinogenesis and the increased rates of lymphoma, The theory of immune surveillance and immunoediting is a dynamic process involving immune recognition and elimination of cancer, an equilibrium state and at times evasion of cancer from immune system control (1-3). Immune system avoidance and escape is now a recognized sarcoma, and cervical cancer in immunocompromised individuals support the notion that immunoediting is essential for cancer suppression in humans (2), (4).

checkpoint receptor of the CD28 receptor family (5). The ligand for the PD-1 receptor, PD-L1, is Under chronic stimulation, T cells lose proliferative and effector function capacity, often due to previously correlated with poor patient prognosis and resistance to treatment in non-small-cell lung cancer, glioblastoma multiforme, and squamous-cell carcinoma of head and neck (6-8)]. signal down-modulation via the increased expression of proteins such as PD-1, an inhibitory Binding of ligand (PD-L1 or PD-L2), often expressed on tumor cells, to PD-1 imparts an inhibitory signal to the T cell, thus down-modulating the anti-tumor T-cell response (9). expressed in a variety of human malignancies, and its high level of expression has been

will likely require combining anti-PD-1 monoclonal antibody (mAb) treatment with conventional convergent aspects of host immunity by employing complementary immunomodulators as well approach to stimulating the immune response, and has achieved significant objective responses as immune-stimulatory aspects of conventional modalities such as radiation and chemotherapy in advanced, melanoma, renal cell cancer (RCC), and NSCLC (10). However, optimal therapy Blockade of the PD-1/PD-L1 T-cell checkpoint pathway is an effective and well tolerated therapies and novel immunotherapy approaches. Combination approaches to stimulate may result in the development of more effective cancer therapies.

## 1.1 RADIATION THERAPY AND IMMUNOGENICITY

outside of a radiation treatment field after radiation therapy. It is thought to be immune mediated "damage-associated molecular patterns" (DAMP's) (14). Chemokines and cytokines such as ILand has sparked interested in multi-modal therapies (11-13). Radiotherapy is known to induce 1B and TNF-A, as well as heat shock protein 70 (HSP70), high mobility group box 1 protein (HMGB1) and adenosine triphosphate (ATP) serve to recruit dendritic cells. Also, DAMP's The abscopal effect is a well described phenomenon in which tumor regression is observed immunogenic cell death in cancer cells, marked by the expression of molecules that elicit

cells show increased expression of tumor specific antigen and antigen-presenting complexes and development of an appropriate adaptive immune response (15, 16). Likewise, radiotherapy has novo transcription and up-regulation of tumor antigen proteins in lung cancer cell lines. These been shown to induce the expression of the antigen-presenting molecule MHC-1 as well as de induce maturation of dendritic cells enabling antigen presentation, and subsequently the demonstrate increased susceptibility to cytotoxic T-cell killing (17).

blocking monoclonal antibody (19). Lee et al. showed that ablative doses of radiation correspond that ablative radiotherapy delivered in a hypofractionated regimen more frequently produces an lymphocytes and reducing immune mediated cancer killing (20). In a pre-clinical mouse model radiation treatment can produce an individualized "in situ vaccine" against the tumor cells that receptors mediating T-cell recognition and killing (18). Pre-clinical studies have demonstrated fractionated radiation therapy impairs immune response due to increased killing of circulating of metastatic breast carcinoma, three doses of 8Gy was superior to a single dose of 20Gy or 5 tumor antigens from killed cells and increasing tumor cell surface expression of antigens and abscopal effect, especially when combined with immunotherapy compared to conventionally to greater levels of dendritic cell maturation and T-cell priming in draining lymph nodes in a Radiation therapy may sensitize tumor cells to immune-mediated attack by releasing soluble mouse model of melanoma (21). Taken together, there is increasing evidence that ablative doses of 6Gy of irradiation in inducing an abscopal effect in mice treated with a CTLA-4 fractionated radiation therapy (19). Researchers have speculated whether conventionally could work in concert with immunotherapy (22-24).

observed in preclinical mouse models as well as in human studies (26, 27). Antigenic cascade has been suggested as an essential component of abscopal tumor regression and that radiation potentially cause polyclonal T-cell responses to a variety of tumor antigens through antigenic cascade leading to a robust immune response against tumor tissues that harbor these antigens particular tumor antigen results in the acquisition of novel tumor antigens and activity of the therapy, by inducing an immunogenic cell death, when coupled with immunotherapy, can immune system toward these newly discovered antigens (25). Antigenic cascade has been "Antigen cascade" is a term used to describe the process in which vaccination against a

T-regulatory (T-reg) cell representation in the tumor microenvironment after radiation therapy is tumor cells (24),(28, 29). However, the increased presence of T-reg cells following SBRT in the any benefit obtained from increased antigen release, enhanced antigen presentation, or influx of The influx of T-reg cells into an irradiated tumor microenvironment therefore may counteract vigorous immune response since T-reg cells promote tolerance of the immune system toward specific immune suppression mediated primarily by T-regs develops over several weeks (18) a known phenomenon (20). Following sublethal irradiation of antigen-primed mice, antigen-T effector cells. This observation is often used to suggest that radiation therapy impedes a

functional analysis of these T-reg cells reveal impairment and inability to prevent T cell tumor microenvironment does not correlate with increased immunosuppression. In fact, proliferation (30).

suppressive responses to conventional fractionated radiation therapy creating a prime opportunity for enhanced tumor response when combining SBRT with immune modulating agents. Given the improved outcomes with immunotherapy relative to cytotoxic chemotherapy, it is plausible that enhanced response with combined modality approaches could yield further improvements in These studies suggest high dose hypofractionated radiation abrogates immune system clinical outcomes.

## 1.2 RATIONALE FOR ANTI-PD1 BLOCKADE.

expression as a mechanism of immune system evasion. Hence, PD-L1 expression by tumor cells upregulating T-reg cells (31). Tumor cells have been shown to upregulate PD-1 ligand (PD-L1) immunotherapy target and has been demonstrated as an effective approach to overcome cancer contributes to immune system evasion by tumors (32). As such, PD-1 blockade is an obvious PD-1 is a cell surface molecule frequently expressed on the surface T-cells. It functions as an immune checkpoint and down regulates the immune system by preventing activation and proliferation of T-cells by increasing programmed cell death in cytotoxic T-cells and mediated immunosuppression.

alone (34). Moreover, up to 40% of mice treated with combination therapy survived longer than glioma, combination radiation therapy and anti-PD-1 blockade resulted in increased number of combined with PD-1 inhibition promoted tumor-associated antigen / MHC complex formation Within the past several years, several groups have employed the use of radiotherapy with PD-1/PD-L1 signaling inhibition in mouse models with remarkable results. Ablative radiotherapy infiltration into tumors in a mouse model of melanoma (33). In a mouse model of intracranial 90 days compared to  $\sim$  30-day survival for either treatment alone and these "cured" mice also killer T-cells and decreased T-reg cell infiltration in tumors when compared to either therapy and subsequent antigen cross-presentation within lymph nodes followed by cytotoxic T-cell developed long-term immunity and were resistant to re-inoculation with tumor cells.

PD-1 expression by tumor cells prevents immune system recognition of distant metastases (35). In this mouse mouse model study of metastatic melanoma, PD-1 inhibition resulted in a 66% reduction in secondary non-irradiated tumors 20 days after a single ablative dose radiation. A single dose of 15Gy was chosen since this therapy is representative of SBRT aimed at controlling oligometastatic disease in humans.

## 2.0 PROPOSED TRIAL RATIONALE

progression on or after platinum based therapy. In the open-label trial, patients were randomized improved to 9.2 months compared to 6 months in patients receiving docetaxel (n=137)  $75 \text{mg/m}^2$ months compared to 2.8 months but 1 year overall survival was improved to 42% compared to approved in February of 2015 by the FDA for patients with metastatic squamous NSCLC with Anti-PD-1 antibodies have demonstrated activity in the treatment of lung cancer. Opdivo was to receive OPDIVO (n=135) administered at 3mg/kg every 2 weeks. Median survival was every 3 weeks, p=0.00025. Median progression free survival was slightly improved to 3.5 24% (36).

free survival and resultant significant increases in overall survival beyond 3 months. We propose effect seen with combined modality treatment will result in improved local control, progression We expect that improvements in local control, increased immunogenic response and abscopal a pilot/phase II study to assess the safety and efficacy of combination immunotherapy and stereotactic ablative radiation therapy (I-SABR).

treatments followed by immunotherapy following the conclusion of SABR/SBRT. This approach presentation and upregulation of PD-1 by tumor cells following ablative radiation therapy. After an interim safety analysis, the study will continue to the phase II portion where overall survival, progression free survival and response rate will be the primary and secondary end points. For Treatment will be a sequential combination treatment of SABR/SBRT and immunotherapy to assess the safety and feasibility of treatment. SABR/SBRT will be administered in 3-5 daily reference, outcomes will be compared to the immunotherapy arms of checkmate 057 and will take advantage of the transient increase in antigen availability, increased antigen Keynote 042 trials.

Several trials examining combination I-SABR are currently underway. A table of selected studies is included in Table 1.

| Study | SABR | Dose | Immunotherapy | Sequence |
|---|---|---|---|---|
| (Institution) | Target | (Gv/Fractionation) | Agent | |
| NCT02239900 | Liver | 50/4 | Ipilimumab | Concurrent/Sequential |
| (MD Anderson | Lung | 60/10 | | |
| Cancer Center) | Adrenal | | | Alegary (Management of the Control o |
| NCT01862900 | Lung | 15/1 | Anti-OX40 | Concurrent |
| (Chiles Research | Liver | 201/1 | | |
| Institute) | | i i i i i i i i i i i i i i i i i i i | | |
| NCT01769222 | Any | 20/2 | Ipilimumab | Concurrent |
| (Stanford University) | | | | |
| NCT02298946 | Liver | 8/1 | PD-1 Inhibitor | Sequential |
| (NIH/NCI) | | 24/3 | | |

Table 1. List of selected ongoing I-SABR studies

## 2.1 RATIONALE FOR DOSE SELECTION

institutional randomized trial from MD Anderson cancer center, patients with oligmetastatic lung explored in multiple studies with encouraging long term survival data (37-39). In a recent multcancer where randomized to systemic therapy plus SBRT to all metastatic sites versus systemic significantly improved in progression free survival in the SBRT group (11.9 vs 3.9 months) at median compared to patients on systemic therapy alone suggesting SBRT acted similarly to systemic A. Radiation Therapy: All patients in this trial will be treated with fractionated Stereotactic therapy alone (40). The study was terminated early after a planned interim safety analysis showed follow up of 12 months. Patients in the SBRT group were less likely to develop new lesions body radiation therapy. Treatment of oligometastatic lung cancer in this fashion has been

prescribed in the NRG-BR001 protocol examining the role of SBRT for oligo-metastatic disease (41). Dose reductions are allowed to pre-specified doses at the treating physician's discretion if fractionated radiation regimens of 8 Gy  $\times$  3 or 6 Gy  $\times$  5 administered on consecutive days, but resulted in abscopal effects. For uniformity, we will adhere to the radiation dose guidelines as dosimetric criteria are not achievable. Dose schedules and prescriptions are described under In a series of mouse tumor models treated with an anti-CTLA-4 antibody combined with 3 not with 20 Gy  $\times$  1 (19). The fractionated regimens, but not the single radiation dose, also different radiation regimens, enhanced tumor responses were observed when treated with radiation treatment.

Pembrolizumab at FDA approved dosing and indications (1, 36). If new FDA approved anti-PDschedules are established and have a favorable toxicity profile and will allow direct comparison allow addition of newly approved therapies to the protocol. (36). These FDA approved dosing 1 therapies emerge during the study duration, the study will be modified with IRB approval to B. Immunotherapy: All patients in this trial will be treated with either Nivolumab or of outcomes to immunotherapy alone trials vs immunotherapy plus SBRT.

### 3. STUDY OBJECTIVES

### 3.1 Primary Objectives

The primary objective of the pilot phase of the study is to characterize the safety, feasibility and tolerability of sequential combination I-SABR in patients with metastatic NSCLC. The first 20 enrollment. In the Brahmer trial, 5% of patients in the Nivolumab arm developed pneumonitis patients will be evaluated for 15 weeks following treatments with I-SABR prior to continuing patient with pulmonary events were treated with glucocorticoids and all cases resolved with a with a median time to onset of treatment related pulmonary events of 15 weeks. All but one median time to resolution of 5 weeks (range 0.6-12.1 weeks). If more than 5% of patients develop grade ≥ 3 pneumonitis during the initial evaluation phase, no lung directed therapy will be permitted during the phase II portion.

The primary objective of the phase II portion of the study will be overall survival.

### 3.2 Secondary Objectives

The secondary objectives of the study are

- To determine the progression free survival measured from time of enrollment to first evidence of progressive disease and evaluated 3 months after treatment initiation.
- progressive disease at the treatment site and evaluated 3 months after treatment initiation To determine the local control measured from time of enrollment to first evidence of તં
  - To determine the incidence of grade  $\geq 3$ , pneumonitis 6 months of completing SBRT
    - To determine the influence of number of metastatic sites on OS, and PFS.

#### 4. STUDY DESIGN

## 4.1 STUDY DESIGN AND DURATION

NSCLC. Treatment safety and feasibility will be assessed in the initial pilot phase and oncologic This is a combination single arm pilot/Phase II study of combination I-SABR for metastatic outcomes will be assessed in the second phase.

After screening, patients will receive 3-5 fractions of SBRT/SABR to up to 3 metastatic sites in addition to the primary tumor. Following the conclusion of SBRT/SABR, patients will receive Immunotherapy therapy at standard dosing until disease progression or discontinuation of treatment due to toxicity or patient choice (Figure 1). Tumor assessment will be performed prior to SABR initiation and every 3 months or for clinical disease progression.

Figure 1: Sample Patient Treatment and Follow-Up Timeline



### 4.2 Radiation Therapy

directed to up to three separate metastatic sites in addition to the primary tumor. Symptomatic or dosimetric criteria cannot be met with stipulated doses, a default dose of 30-40 Gy in 5 fractions at risk disease sites should be prioritized. Strict adherence to dosimetric criteria is required. If Radiation therapy will be delivered using SABR or SBRT using the CyberKnife radiosurgery system. Treatment will be delivered in 3-5 fractions as specified in Table 2. SBRT can be delivered to the PTV to satisfy protocol constraints. 90% will be considered an acceptable will be prescribed. In all cases, a minimum dose of 95% of the prescribed dose is must be minimal deviation.

#### 4.3 Immunotherapy

1/PD-L1 agents. Dose reductions are appropriate for toxicity as specified or at the discretion of Immunotherapy will be delivered in the form of PD-1/PD-L1 blockade using approved anti PD the treating medical oncologist. Prior immunotherapy as part of multi-drug therapy or monotherapy is acceptable prior to initiation of SBRT. The DLT observation period for continuation or discontinuation of therapy is defined as 14 days Any of the below outlined events occurring during each DLT observation period and considered starting with cycle 1, day 1. To be evaluable for DLT, a patient must have received at least the first 2 administrations and be monitored for at least 14 days following the first administration. to be at least possibly related to Nivolumab will qualify as a DLT.

## Non-Hematologic Toxicity

- Grade ≥2 uveitis
- 2. Any Grade ≥3 non-hematologic toxicity except
- a. Nausea, vomiting or diarrhea
- o. Clinically insignificant laboratory abnormalities
- Grade 3 infusion reactions that respond to medical management
- Grade 3 immune related effects other than uveitis that improve within 7-14 days with steroid treatment (Appendix 1)

#### Hematologic Toxicity

- .. Grade 4 neutropenia lasting more than 1 week
- 2. Grade 4 thrombocytopenia
- . Grade 3 thrombocytopenia with bleeding
- Grade ≥3 febrile neutropenia

#### Special

1. Grade  $\geq 2$  pneumonitis

#### 4.4 Duration of Study

short overall survival in patients with metastatic NSCLC, all end-points should be realized within 24 months. At the conclusion of the study, patients and investigators may decide to continue with The study will conclude 24 months after the last patient is accrued. Given the poor prognosis and Immunotherapy treatment. We expect to enroll 100 patients over 2 years.

## 5. PATIENT ELIGIBILITY AND CRITERIA

The target study population comprises patients with metastatic lung cancer who are eligible for an immunotherapy agent as monotherapy or combination therapy.

#### 5.1 Inclusion Criteria

- 1. Histologically or cytologically confirmed Stage IV NSCLC according to the 7th AJCC staging manual. Patients with recurrent disease after definitive treatment with surgery or concurrent chemoradiation are eligible.
- immunotherapy or single agent monotherapy are eligible. Patients who progress on maintenance immunotherapy are eligible if sites of progression are amenable to local therapy for control. 2. Patients must be eligible for an immunotherapy agent as determined by treating medical oncologist. Patients who progress after drug therapy (3 months) for ALK, EGFR or ROS mutation positive lung cancer are eligible. Patients who received prior combination
- 3. At least 2 lesions that are safely amenable to SBRT/SABR.
- 4. ECOG ≥2.
- (RECIST) 1.1 criteria for response assessment or at least 1 lesion with FDG avidity and CT 5. At least 1 measurable lesion according to Response Evaluation Criteria in Solid Tumors correlate that can be monitored for PET-CT response by SUV Max increase or decrease.
- $6. \ge 18$  years old.
- 7. Normal Hepatic and renal function.
- 8. Bone marrow reserve:
- a. ANC  $\ge 1.5 \times 10^9 / L$
- b. Hemoglobin ≥9.0 g/dL
- c. Platelet count  $\geq$ 75 x 10 $^9$ /L
- 9. Ability to comply with follow-up visits and evaluations, treatment planning and studies and other study related procedures and visits.
- 10. Ability to sign informed consent.

### 5.2 Exclusion Criteria

1. Patients with active CNS metastases. If metastases are treated and patients return to baseline and no steroids are required, patients are eligible. 17-009 11 PCK-01

- 2. Active, known or suspected auto-immune disease.
- 3. Patients with medical conditions that require systemic immunosuppression.
- 4. Patients with a history of interstitial lung disease.
- 5. Other active malignancy requiring intervention.
- 6. Prior lung radiation, with the only metastatic targets in the lungs.
- 7. Unresolved toxicity from prior chemotherapy or anti-cancer treatment.
- 8. Current or prior enrollment in clinical trial with an investigational drug within 4 weeks.
- 9. Pregnancy or positive pregnancy test.

#### 5.3 Sample Size

More than 350 patients with metastatic lung cancer present to the Crozer-Keystone health system feasibility analysis will be performed on the first 20 patients in the pilot phase. Overall survival, 100 patients will enroll and be treated on this study. Patients will be followed for 2 years on the for treatment annually. If 50% of patients are eligible for this study, we expect approximately progression free survival, local control and subgroup analysis will be performed on the entire study. The study will conclude 2 years after the last patient is enrolled. An interim safety and patient cohort at the conclusion of the study.

## 5.4 Discontinuation of Study Treatment

Patients who discontinue study treatment will be asked to return to the clinic for all remaining study visits per the visit schedule, and will be expected to continue with relevant study assessments.

## 5.5 Withdrawal from Study

During the treatment period and follow-up period, a patient who withdraws consent to continue participation in the study will be removed from follow-up requirements. Routine clinical care will continue but no data will be collected for study purposes.

## 6. RADIATION THERAPY

## 6.1 Specifications for Radiation Therapy

specified in Table 2 for a given treatment site. Treatment at the protocol defined dosing regimen 95% of the prescribed dose must be delivered to the treatment planning volume (PTV). 90% will is only permitted if the normal tissue criteria are met. As a default dosing scheme, if dosimetric criteria are not achieved, then a dose of 30 Gy in 5 fractions will be delivered. A minimum of primary lung tumor may be treated as well. Patients will receive the radiation therapy dose SBRT/SABR will be delivered to up to three separate metastatic sites in 3-5 fractions. The be considered an acceptable minor deviation.

irradiation while sparing normal tissue in accordance with standard radiation oncology practice. If symptomatic or at risk lesions are present, these lesions should be prioritized for the target The lesions selected for treatment should be lesions that can be safely irradiated with focal selection. No more than one lung lesion may be treated.

Table 2. Specified SBRT/SABR Prescription Doses

| Lesion Location | Dose/Fractionation | Acceptable Variation |
|---|---|---|
| Lung-Peripheral Lesion | 45 Gy/3 fractions | 40 Gy/5 fractions |
| Lung-Central Lesion | 50 Gy/5 fractions | 40 Gy/5 fractions |
| Mediastinal/Cervical Node | 50 Gy/5 fractions | 40 Gy/5 fractions |
| Liver | 45 Gy/3 fractions | 40 Gy/5 fractions |
| Spine/Para-spinal | 30 Gy/3 fractions | 30 Gy/5 fractions |
| Bone (Other than spine) | 30 Gy/3 fractions | 30 Gy/5 fractions |
| Adrenal Gland/Pelvic Metastases 45 Gy/ 3 fractions | 45 Gy/ 3 fractions | 40 Gy/5 fractions |

## 6.2 Radiation Therapy Simulation

for the potential for respiratory motion. Daily IGRT with CBCT is required for all treatment sites required for tumor tracking. Respiratory motion management (RMM) is required for all lesions required for central lung lesions and liver metastases. For other sites, the use of IV contrast is All patients will undergo immobilized 1mm CT scans for treatment planning. IV contrast is encouraged and left to the discretion of the treating radiation oncologist. Fiducials may be when an approved non-CyberKnife treatment system is utilized.

## 6.3 Treatment Planning and Target Volumes

Location: Each lesion will be assigned to one of the 7 locations specified in Table 2

Lung Peripheral Lesion: The lesion is outside the proximal bronchial tree as defined as within 2cm in all directions around the carina, right and left main bronchi, right and left upper lobe bronchi, intermedius bronchus, right middle lobe bronchus, lingular bronchus and right lower lobe bronchi. The lesion does not the mediastinal or pericardial pleura.

Lung Central: The lesion is within 2cm of the proximal bronchial tree.

Mediastinal/Cervical Node: The lesion arises in the anatomic mediastinum or cervical lymph node levels I-VI or retropharyngeal space.

Liver: Lesion is located inside or touches the liver parenchyma.

Spine or Paraspinal: Lesion is located within vertebral body or within 1cm of a vertebral body, pedicle or posterior elements.

**Bone:** Lesion is located within a bony structure (excluding spine).

Adrenal Gland/Pelvic Metastases: Lesion arises within the adrenal gland or within the true pelvis or inguinal nodes.

## 6.4 Target Delineation and Treatment Planning

The gross tumor volume (GTV) will be contoured in the appropriate CT window. Rigid PET-CT/MRI fusion is allowed to assist in target delineation when necessary

No clinical target volume (CTV) expansion is allowed. GTV=CTV.

for motion susceptible targets. The expiratory and inspiratory phase scans (Phase 0 and 50) from caution because lung and MIP reconstructions may erroneously generate an ITV when breathing For non-fiducial based tracking treatments, an internal target volume (ITV) must be generated a 4D-CT are suggested for defining the ITV. MIP reconstructed images should be used with is irregular or when lesions abut soft tissue structures.

A 3-5mm uniform expansion will be added to generate the planning target volume (PTV).

95% of the prescribed dose should encompass 100% of the PTV.

### 6.5 Organs at Risk (OAR)

OAR must be contoured. The specific OAR to be contoured will depend on the location of lesion being treated

# Lung Central/Lung Peripheral/Mediastinal/Cervical Lymph Node metastases:

The proximal tracheobronchial tree, lungs, left/right/combined, heart, esophagus, spinal cord, chest wall, brachial plexus (when at risk), skin, liver, larynx, stomach will be contoured.

## Abdominal-pelvic metastases (liver, adrenal, lymph nodes):

The stomach, duodenum, spinal cord, kidneys, large and small bowel, rectum, bladder, lungs, and cauda will be contoured.

#### Spinal Metastases:

guidelines for target delineation. A partial spinal cord volume 6mm above and below the target All spine target volumes will be contoured per the international spine radiosurgery consensus region will be contoured. Additional OAR will be based on the spine level.

## 6.6 Dose Limits and DVH Criteria

#### See Appendix II.

## 6.7 Evaluation of Targeted Lesions

Targeted lesions will be evaluated on 3 month interval scans or scans procured for clinical progression. Evaluated lesions will be described as follows:

Complete Response (CR): Disappearance of target lesion.

Partial Response (PR): At least 30% decrease in the sum of the diameters of the target lesions using the baseline sum of diameters.

smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an **Progressive Disease (PD):** At least 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the absolute increase of at least 5 mm (0.5 cm).

Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.

6.8 Evaluation of Non-Target Lesions

Complete Response (CR): Disappearance of all non-target lesions and normalization of tumor All lymph nodes must be non-pathological in size (<10 mm [<1 cm] short axis).

Progressive Disease (PD): Unequivocal progression of existing non-target lesions. It must be representative of overall disease status change, not a single lesion increase in size.

### 7. IMMUNOTHERAPY

Immunotherapy administration will commence or continue following the conclusion of SBRT/SABR

as an IV push or bolus injection. At the end of the infusion the administration line will be flushed Immunotherapy will be administered as an IV infusion as specified. It is not to be administered with a sufficient quantity of normal saline per standard of care. Infusions will continue on a standard schedule for the specific immunotherapy agent with pre-treatment assessments for adverse effects using a standard questionnaire.

Immunotherapy administration will be delayed in the case of any of the following:

Any Grade ≥ 2 non-skin, drug-related adverse event, with the following exceptions:—Grade 2 drug-related fatigue or laboratory abnormalities do not require a treatment delay

Any Grade 3 skin, drug-related adverse event

Any Grade 3 drug-related laboratory abnormality, with the following exceptions for lymphopenia, leukopenia, AST, ALT, or total bilirubin:

- Grade 3 lymphopenia or leukopenia does not require dose delay
- If a subject has a baseline AST, ALT or total bilirubin that is within normal limits, delay dosing for drug-related Grade≥2 toxicity
- If a subject has baseline AST, ALT, or total bilirubin within the Grade 1 toxicity range, delay dosing for drug-related Grade  $\geq 3$  toxicity

Any adverse event, laboratory abnormality, or intercurrent illness which, in the judgment of the investigator, warrants delaying immunotherapy administration.

## 7.1 Dose reductions and modifications

There will be no dose reduction or modifications in Immunotherapy administration.

## 7.2 Treatment Compliance

Treatment compliance will be monitored by the site P.I and documented in the medical record

## 8.0 PATIENT ASSESSMENTS

#### 8.1 Study Parameters

See Appendix III

#### 8.2 Data Collection

Patients will be stratified by number of metastatic lesions. <3 lesions, 4-5 lesions and >5 lesions.

All study data will be coded and de-identified. Codes and patient data will be stored separately in a password protected file. Any hard copies will be stored in a locked file cabinet. All other data will be stored on a password secured and encrypted computer only accessible to study staff.

Adverse event data collection and reporting, which are required as part of every clinical trial, are future studies using similar agents. Adverse events are reported in a routine manner at scheduled done to ensure the safety of patients enrolled in the studies as well as those who will enroll in times during the trial by the study investigator.

For pre-specified time points and required reporting please see Appendix IV.

## SUPPORTIVE CARE GUIDELINES FOR SPECIFIC DRUG-RELATED ADVERSE EVENTS APPENDIX I. RECOMMENDED DOSE MODIFICATION OR DISCONTINUATION AND

| | CTCAR | Wanagement | | | Differential |
|---|---|---|---|---|---|
| | v4.03 | Managomone | | ſ | |
| Event(s) | Grade | | Action/Supportive Care Guidelines | Symptomsa | Diagnosis |
| Colitis events | ≤ Grade | No change in dose | For diarrhea, treat symptomatically (loperamide, oral hydration, electrolyte | Symptoms<br>may | All attempts |
| bowel • obstruction | | | substitution and ALA collins diety. Endoscopy is recommended if symptoms | mclude (but | should be made |
| <ul> <li>Colitis</li> </ul> | | | persist. | not limited to): | to rule out other |
| • Colitis | | | <ul> <li>Grade 1 diatrica that persist for &gt;1 week<br/>should be treated with the addition</li> </ul> | Abdominal | causes such as |
| microscopic | | | of oral diphenoxylate hydrochloride and atropine sulfate four times daily and | pain,<br>cramping | metastatic |
| | | | budesonide 9 mg daily. | and/or<br>bloating | disease, bacterial |
| Enterocolitis | Grade 2 | Hold until ≤Grade<br>1. | GI consultation and endoscopy is recommended to confirm or rule out colitis | Blood and/or | or parasitic |
| | | ŗ | for grade 2 diarrhea that persists >1 week or | mucus in | |
| hemorrhagic | | Kesume at same | grade 1-2 diarrhea with rectal<br>bleeding (additional guidelines for the | stool<br>with or | infection, viral |
| Gastrointestinal | | dose level. May | treatment of persistent colitis are | without | gastroenteritis, |
| (GI) perforation | | increase dosing | provided below). | fever | or the first |
| Necrotizing | | if | addition of oral diphenoxylate | <ul> <li>Constipation</li> </ul> | manifestation of |
| • | | | hydrochloride and atropine sulfate four | • | |
| colitis<br>Diambea: | | it takes more than | times daily and budesonide 9 mg | Diarrhea Hens | an inflammatory<br>bowel disease by |
| , 101 110a. | | toxicities to | Grade 2 diarrhea with diffuse ulceration and | Nausea | |
| tients who | | resolve. | bleeding seen on endoscopy | • and/or | examination for |
| , | | | may require oral steroids with prolonged | | stool teahouytes, |
| experience diarrhea | | | taper and represent an increased risk for the development of bowel perforation. | Vomimig | stool cultures, |
| should be advised to | | | Consider prophylactic antibiotics | • Peritoneal | |
| drink liberal | | | for opportunistic infections. | signs | and a<br>Clostridium |
| | | | When symptoms improve to Grade 1 or less, | consistent | |
| quantities of clear<br>fluids. If sufficient | | | statorid taper should be statted and continued over no less than 4 weeks. | bowel | difficile titer. |
| | | | • In patients with Grade 2 enterocolitis, | | |
| | | | IMMUNOTHERAPY should be withheld | 3 | |
| oral fluid intake is | | | and<br>antidiarrheal treatment should be ctarted. If | perforation <br> Rectal | |
| not feasible, fluid | | | symptoms are persistent for | • bleeding | |
| | | | more than one week, systemic | ) | |
| and electrolytes | | | corticosteroids should be initiated (eg, | With or | |
| should be | | | When symptoms improve to | without fever | |
| | | | Grade 1 or less, corticosteroid taper should | | |
| substituted via IV | | | be started and continued over at | Patients with | |
| infusion | | | least 1 month. | be | |

| | ,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,, | | - Later and the second |
|---|---|---|---|
| | CTCAE | Management | |
| Event(s) | v4.03 Grade | ··· | Action/Supportive Care Guidelines |
| Colitis events | Grade 3-4 | Withhold IMMUNOTHER AP | • In patients with Grade 3 enterocolitis, OPDIVO will be permanently |
| (continued) | | Y | discontinued and treatment with systemic corticosteroids should be initiated |
| | | | at a dose of 1-2 mg/kg/day of prednisone or equivalent. When symptoms |
| | | Discontinue if | improve to Grade 1 or less, corticosteroid taper should be started and |
| | | corticosteroid dose | continued over at reast 1 month. Consider propayated antibroades for opportunistic infections. |
| | | to < 10 mg per day | |
| | | prednisone | For Grade 3-4 diarrhea (or Grade 2 diarrhea that persists after initial steroid |
| | | equivalent within | treatment), |
| | | 12 weeks of toxicity | <ul> <li>Rule out bowel perforation. Imaging with plain films or computed</li> </ul> |
| | | | tomography (CT) can be useful. |
| | | | <ul> <li>Consider consultation with gastroenterologist and confirmation biopsy with</li> </ul> |
| | | | endoscopy. |
| | | | <ul> <li>Treat with intravenous (IV) steroids (methylprednisolone 125 mg) followed</li> </ul> |
| | | | by high-dose oral steroids (prednisone 1-2 mg/kg once per day or |
| | | | dexamethasone 4 mg every 4 hours). When symptoms improve to Grade 1 or |
| | | | less, steroid taper should be started and continued over no less than 4 weeks. |
| | | | Taper over 6-8 weeks in patients with diffuse and severe ulceration and/or |
| | | | bleeding. |
| | | | <ul> <li>If IV steroids followed by high-dose oral steroids does not reduce initial</li> </ul> |
| | | | symptoms within 48-72 hours, consider treatment with infliximab at 5 mg/kg |
| | | | once every 2 weeks. Discontinue infliximab upon symptom relief and |
| | | | initiate a prolonged steroid taper over 45–60 days. If symptoms worsen |
| | | | during steroid reduction, initiate a retapering of steroids starting at a higher |
| | | | dose of 80 or 100 mg followed by a more prolonged taper and administer |
| <u> </u> | | | infliximab. CAUTION: infliximab is contraindicated in patients with bowel |
| | | | perforation or sepsis. |
| *************************************** | | | <ul> <li>If symptoms persist despite the above treatment a surgical consult should be</li> </ul> |
| | | | obtained. |

| January, | | | Addition of the second of the | | |
|---|---|---|---|---|---|
| | CTCAE | Management | | | Differential |
| Event(s) | v4.05<br>Grade | | Action/Supportive Care Guidelines | Symptoms <sup>a</sup> | Diagnosis |
| Endocrine events | Grade<br>1-2 | No change in<br>dose | Monitor thyroid function or other hormonal<br>level tests and serum chemistries<br>more frequently until returned to baseline | Symptoms may | All attempts |
| Hyperthyroidism Hypophysitis Hypopituitarism | а | | values. | include (but not limited to): • Abdominal | should be made<br>to rule out other<br>causes such as |
| Endocrine events | Grade<br>3-4 | Hold until on stable | • Consider endocrine consultation. | pain | brain metastases, |
| Hypothyroidism | | replacement dose | <ul> <li>Rule out infection and sepsis with appropriate<br/>cultures and imaging.</li> <li>Replacement of appropriate hormones as</li> </ul> | Abnormal thyroid | sepsis, and/or<br>infection. An |
| Thyroid disorder Thyroiditis | <del></del> | | required. | function tests | endocrinology<br>consultation is |
| Endocrine events | Grade<br>1-4 | Hold until on stable | <ul> <li>Thyroid hormone and/or steroid replacement<br/>therapy to manage adrenal</li> </ul> | chemistries | recommended |
| Adrenal | | replacement dose | insufficiency. If Grade 1—2 hypophysitis is considered. | (Thyroid- | |
| insufficiency | | | pituitary gland imaging should be considered (magnetic resonance imaging | stimulating | |
| Hypophysitis | | | [MRIS] with gadolinium and selective cuts of the nitritary can show | hormone | |
| • Pan- | | | enlargement or heterogeneity and | increased | |
| hypopituitarism | | | confirm the diagnosis). | [decreased], | |
| : 1<br>: 1 | | | ノ <u>ら</u> り | thyroxine | |
| | | | hypotension, dehydration, and electrolyte abnormalities (such as | increased,<br>Tri- | |
| | | | hyponatremia and hyperkalemia) constitutes adrenal crisis. Hospitalization | iodothyronin<br>e | |
| | | | and IV methylprednisolone should be | increased.) | |
| | | | יוורת פיייסיי | Arrhythmias <sup>c</sup> | |
| | | | | intolerance<br>Fatione | |
| | | | | Hypotension <sup>c</sup> | |
| | | | | • Loss of | |
| | | | | appetite • Mental status | |
| | | | | and/or<br>behavior | |
| | | | | changes | |
| | | | | Nausea<br>• and/or | ٠ |
| | | | | Unusual • bowel | |
| | | | | Vision disturbances | |

| 100 Miles | CTCAE | Management | | | Differential |
|---|---|---|---|---|---|
| F | v4.03 | | | Cymptome | |
| Event(s) | Grade | | ┪ | Symptoms | Diagnosis |
| Eve event | Grade 1 | Discontinue | <ul> <li>Evaluation by an ophthalmologist is strongly recommended</li> </ul> | Symptoms | All attemnts |
| | 2 | IMMUNOTHERAPY | pical steroids such as 1% | include (but | |
| Uveitis | | Ħ | | are | should be made |
| | | | | not limited | |
| (iritis, iridocyclitis) | | symptoms persist | iridocyclitics. | to): | to rule out other |
| | | • | | Blurred | |
| | | despite treatment | | • vision | causes such as |
| | | with topical | | <ul> <li>Diffuse</li> </ul> | metastatic |
| | | • | | erythema | |
| | | immunosuppressive | | and a | disease, |
| | | therapy | | prominent | infection, or |
| | ر جامين | مانون | <ul> <li>Evaluation by an ophthalmologist is strongly</li> </ul> | blush on the other ocular | other ocular |
| | | HERAPY | • Treat with topical steroids such as 1% | | |
| | | if | prednisolone acetate suspension and | sclerae | disease (e.g., |
| | | | • | Dryness of | 1 |
| | | symptoms persist | iridocyclitics. | • the | glaucoma or |
| | | despite treatment | | eyes | cataracts). |
| | | with topical | | • Pain | |
| | | immunosuppressive | | <ul> <li>Photophobia</li> </ul> | |
| | | therapy and do not | | | |
| | | improve to Grade 1 | | | |
| | | within the | | | |
| | | retreatment period | | | |
| | | OR requires | | | |
| , michael | | systemic treatment. | | | |
| | Grade 3- | - | <ul> <li>Treat with systemic corticosteroids such as</li> </ul> | | |
| | 4 | Discontinue | prednisone at a dose of | | |
| | | | 1-2 mg/kg per day. When symptoms | | |
| | | IMMUNOTHERAPY. | improve to ≤Grade 1, steroid taper | | |
| | | | should be started and continued over no less | | |
| | | | than 4 weeks. | | |

| | CTCAE | CTCAE Management | | | Differential |
|---|---|---|---|---|---|
| Event(s) | v4.03<br>Grade | | Action/Supportive Care Guidelines | Symptoms <sup>a</sup> | Diagnosis |
| Hepatic events | Grade 1–2 Withhold | Withhold | <ul> <li>Monitor liver function tests more frequently<br/>until returned to baseline values.</li> </ul> | Symptoms<br>may | All attempts |
| Usnotitie | | IMMUNOTHERAPY | | include (but<br>are | should be made |
| Hepatitis, | | is a treatment- | | not limited to): | not limited to): to rule out other |
| • | | | | Elevations | |
| Autoimmune | | emergent concurrent | | • in: | causes such as |
| | | elevation of ALT | | )<br>X | metastatic |
| | | and bilirubin that | | ULN | disease, |
| | | | | o ALT>2.5 | |
| | | corresponds to an | | ×<br>14.11.1 | progressive liver |
| | | upward shift of 2 of<br>more grades in both | | o Total | hepatitis, |
| | | parameters. | | bilirubin<br>>1.5 | alternative drug |
| | Grade 3-4 | Grade 3-4 Discontinue | <ul> <li>Consider appropriate consultation and liver<br/>biopsy to establish etiology of</li> </ul> | × CLN | toxicity, |
| | | IMMUNOTHERAPY | | | |
| | | when | hepatic injury, if necessary. | • Fever | infectious causes |
| | | | <ul> <li>Treat with high-dose IV glucocorticosteroids</li> </ul> | | ; |
| | | AST or ALT | for 24-48 hours. When | Malaise | and/or myositis. |
| | | | symptoms improve to grade 1 or less, a | Upper | |
| | | >5.0 times ULN | steroid taper with dexamethasone | • quadrant | |
| | | ; | 4 mg every 4 hours or prednisone at 1–2 | abdominal | |
| | | and/or total bilirubin | mg/kg should be started and | pain | |
| | | >3.0 times ULN. | continued over no less than 4 weeks. | | |
| - | | | <ul> <li>If serum transaminase levels do not decrease 46</li> <li>hours after initiation of</li> </ul> | | |
| , and delivery | | | systemic steroids, oral mycophenolate mofetil | | |
| | | | 500 mg every 12 hours may | | |
| | | | be given. Infliximab is not recommended due | | |
| | | | to its potential for | | |
| | | | hepatotoxicity | | |
| | | | <ul> <li>Several courses of steroid tapering may be</li> </ul> | | |
| | | | necessary as symptoms may | | |
| | | | worsen when the steroid dose is decreased. | | |

CTCAE | Management |

Differential

Symptoms

| i. | v4.03 | | | |
|---|---|---|---|---|
| Event(s) | Grade | | Action/Supportive Care Guidelines | Diagnosis |
| of White | | No change in | | |
| Neutropenia | ≤Grade 1 dose | dose | | |
| • | | No change in | | |
| | Grade 2 dose | dose | | |
| | | No change in | | |
| | Grade 3 dose | dose | | |
| | | Hold until | | |
| | Grade 4 | resolves | | |
| | | to ≤Grade 1. May | | |
| | | increase the | | |
| | | dosing | | |
| | | interval by 1 | | |
| | | week. | | |
| | | Discontinue if | | |
| | | toxicities do not | | |
| | | resolve within | | |
| | | 12 weeks. | The state of the s | |

| | CTCAE | Management | | | Differential |
|---|---|---|---|---|---|
| Event(s) | Grade | | Action/Supportive Care Guidelines | Symptoms | Diagnosis |
| Pneumonitis events | Grade<br>1 | Consider hold of | • Radiologic findings should be followed on serial Symptoms imaging studies at least | Symptoms<br>may | All attempts |
| Pneumonitis | | therapy. IMMUNOTHERAPY | every 3 weeks. | include (but<br>are | should be made |
| Interstitial | | | | not limited | |
| gunl | | may be continued | <ul> <li>Monitor for symptoms every 23 days.</li> <li>Consider pulmonary consultation and/or</li> </ul> | :(oı | to rule our ouner |
| disease | | with close | bronchoscopy if clinically | Abnormal breath | causes such as |
| Acute interstitial pneumonitis | | monitoring. | indicated. | sounds Chest pain | metastatic<br>disease, bacterial |
| | Grade<br>2 | Hold<br>IMMUNOTHERAPY | To rule out other causes such as infection: | and/or | or viral |
| | : | | <ul> <li>Consider pulmonary consultation with</li> </ul> | c | : |
| | | | bronchoscopy and | tightness | infection. |
| | | | biopsy/bronchoalveolar lavage (BAL). | • Dyspnea | |
| | | | <ul> <li>Consider pulmonary function tests.</li> </ul> | Dry cough | |
| | | | <ul> <li>Follow radiologic findings on serial imaging</li> </ul> | į. | |
| | | | studies every 1-3 days | • rangue | A CONTRACTOR . |
| | | | If the patient is determined to have study drug | £ | |
| | | | associated pneumonitis: | • rever | |
| | | | <ul> <li>Monitor symptoms daily; consider</li> </ul> | | |
| | | | hospitalization. | <ul> <li>Hemoptysis</li> </ul> | |
| | | | <ul> <li>Treat with systemic corticosteroids at a dose of</li> </ul> | | |
| | | | 1–2 mg/kg/day prednisone or | | |
| | | | 1 or less steroid taner should | | |
| | | | be started and continued over no less than 4 | | |
| | | | weeks. | | |
| | | | <ul> <li>Treatment with IMMUNOTHERAPY may be</li> </ul> | | |
| | | | resumed if the event improves to | | |
| | | | Scrade 1 within 12 weeks and corticosteroids | | |
| | | | have been reduced to the | | |
| | | | equivalent of memoriphecursorone to mg of month daily or less Reneat | | |
| : | | | chest imaging monthly as clinically indicated. | | |
| or and a second | ········· | | For Grade 2 pneumonitis that improves to | | |

| | | | | | | | | | | ••••• | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| <ul> <li>≤Grade 1 within 12 weeks, the following rules should apply: <ul> <li>First episode of pneumonitis: May increase dosing interval by one week in subsequent cycles.</li> <li>Second episode of pneumonitis: Discontinue IMMUNOTHERAPY if upon rechallenge the patient develops a second episode of ≥ Grade 2 pneumonitis.</li> </ul> </li> </ul> | Consider pulmonary function tests with pulmonary consult. Bronchoscopy with biopsy and/or BAL is | <ul> <li>Treat with IV steroids (2-4 mg/kg per day<br/>prednisone or equivalent). When</li> </ul> | symptoms improve to grade 1 or less, a high-<br>dose oral steroid (1-2 mg/kg | prednisone once per day or 4 mg dexamethasone every 4 hours) taper should | be started and continued over no less than 4 | weeks. • Add prophylactic antibiotics for opportunistic | infections. | <ul> <li>II IV steroids followed by high-dose oral<br/>steroids does not reduce initial</li> </ul> | symptoms within 48–72 hours, treat with | infliximab at 5 mg/kg once every 2 weeks. Discontinue infliximab upon | symptom relief and initiate a | prolonged steroid taper over 45–60 days. It symptoms worsen during steroid | reduction, initiate a retapering of steroids | starting at a figher dose of 80 or 100 mg followed by a more prolonged taper | and administer infliximab. |
| | Discontinue pulmonary cor • Bronchoscog | IMINIONO I FIENCAL I . | | | | | | | | | | | | | |
| | Grade<br>3-4 | | | | | | | | | | | | | | |
| ; ) | | | | | | | | | | | | ٠ | | | |

| | T | | | | | | | | | | | | | | | | | _ | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Diagnosis | All attempts | should be made | to rule out other | causes such as | uropathy. | progression of | disease or initro | f militar to samana | to other | | chemotherapy | agonts. A renai | consultation is | recommended | | | | | | | | | | | | |
| | Symptoms<br>may | not<br>not | limited to): | <ul> <li>Fatigue</li> <li>High blood</li> </ul> | pressure | • Increased | Senim | | creatinine | | <ul> <li>Swelling</li> </ul> | | | | | *** | | | | | | Tu-th | ••• | | | - |
| Action/Supportive Care Guidelines | Provide symptomatic treatment. Monitor greating weekly | <ul> <li>Monto creamine weekly, when it returns to</li> <li>baseline, resume routine</li> </ul> | creatinine monitoring per protocol. | | | Systemic corticosteroids at a dose of 1-2 • mg/kg/day of prednisone or | equivalent may be indicated. When symptoms improve to Grade 1 or less. | corticosteroid taper should be started and | continued over at least 1 month. | Consider prophylactic antibiotics for | | | • Grade 4. | Renal consultation with consideration of ultrasound and/or hionsy as | appropriate. | <ul> <li>Monitor creatinine daily.</li> </ul> | <ul> <li>Treat with systemic corticosteroids at a dose of</li> </ul> | 1–2 mg/kg prednisone or | <ul> <li>When symptoms improve to grade 1 or less</li> </ul> | steroid taper should be started | and continued over no less than 4 weeks. | Discontinue IMMUNOTHERAPY if unable to | reduce corticosteroid dose for irAEs to | \$10 mg. IMMATNOTHER ARV treatment many be | restarted and the dose modified as specified in | |
| | Consider | withholding | if event | does not improve with symptomatic | treatment | Consider | withholding | ) | IMMUNOTHERAPY. | | | | | Discontinue | IMMUNOTHERAPY. | | | | | | | | | | *** | |
| v4.03<br>Grade | Grade 1 | | | | | Grade 2 | | | | | | | | Grade 3- | | | | | | | | | | | | |
| Event(s) | ents | Nephritis | Nephritis | autoimmune | , | Renal<br>failure | | | | | | | | • | Acute | | | | | | | | | | | _ |
| ( )<br>( ) | Renal ev | • | • | | | • | | | | | | | | • | | | | | | | ) | | | · | | |
| | v4.03 Grade Action/Supportive Care Guidelines | Event(s) Grade Action/Supportive Care Guidelines Symptoms all events Grade 1 Consider Marity Consider Marity Care Guidelines Symptoms may a may | V4.03 Grade Action/Supportive Care Guidelines Symptoms | v4.03 Action/Supportive Care Guidelines Symptoms Grade 1 Consider Provide symptomatic treatment. Symptoms dephritis withholding baseline, resume routine include (but include (but include)) dephritis if event creatinine monitoring per protocol. limited to): | v4.03 Action/Supportive Care Guidelines Symptoms Grade I Consider Provide symptomatic treatment. Imay include (but include (but include)): Vephritis IMMUNOTHERAPY if event does not improve with symptomatic creatinine monitoring per protocol. limited to): vith symptomatic e High blood | v4.03 Action/Supportive Care Guidelines Symptoms Grade 1 Consider • Provide symptomatic treatment. Symptoms lephritis withholding • baseline, resume routine not lephritis if event creatinine monitoring per protocol. limited to): does not improve with symptomatic • Fatigue with symptomatic • High blood treatment • High blood | Event(s) Grade Action/Supportive Care Guidelines Symptoms Lenal events Grade 1 Consider Provide symptomatic treatment. Symptoms Nephritis withholding - baseline, resume routine not not Nephritis if event creatinine monitoring per protocol. limited to): autoimmune does not improve with symptomatic - Fatigue with symptomatic treatment Systemic corticosteroids at a dose of 1-2 Renal Grade 2 Consider - mg/kg/day of prednisone or | Event(s) Grade Action/Supportive Care Guidelines Symptoms Lenal events Grade 1 Consider Provide symptomatic treatment. Symptoms Nephritis withholding - baseline, resume routine not not Nephritis if event creatinine monitoring per protocol. limited to): Autoimmune with symptomatic reatment - Fatigue With symptomatic reatment Systemic corticosteroids at a dose of 1-2 - High blood Renal Grade 2 Consider - mg/kg/day of preduisone or equivalent may be indicated. When symptoms - Increased withholding improve to Grade 1 or less. - Increased | Event(s) Grade Action/Supportive Care Guidelines Symptoms Lenal events Grade 1 Consider Provide symptomatic treatment. Symptoms Nephritis withholding - baseline, resume routine not not Nephritis If event creatinine monitoring per protocol. limited to): - Fatigue Action/Supportive Care Guidelines not not not Momitor creatinine weekly; when it returns to include (but | Event(s) Grade Consider Action/Supportive Care Guidelines Symptoms Renal events Grade 1 Consider Provide symptomatic treatment. Imagy Nephritis withholding - Provide symptomatic treatment. Incention monitoring per protocol. Include (but include (but in | Event(s) Grade Action/Supportive Care Guidelines Symptoms tenal events Grade 1 Consider • Provide symptomatic treatment. Include (but may) Nephritis Withholding • Provide symptomatic treatment. Include (but may) Nephritis If event foots not improve autoimmune Creatinine monitoring per protocol. Imited to): Renal failure Grade 2 Consider • Systemic conticosteroids at a dose of 1-2 or light blood preduisone or equivalent may be indicated. When symptoms improve to Grade 1 or less, continued over at least 1 month. • Increased continued over at least 1 month. Renal failure IMMUNOTHERAPY. Consider prophylactic antibiotics for • Increased creatinine continued over at least 1 month. | Event(s) Grade Consider Provide symptomatic treatment. Symptoms Renal autoimmune Renal failure Grade 2 Consider Provide symptomatic treatment. Provide symptomatic treatment. Imited (but include (b | Event(s) Grade I Consider Provide symptomatic treatment. Symptoms Nephritis Mitholding • Provide symptomatic treatment. Imay Nephritis Mitholding • baseline, resume routine Incention or creatinine weekly; when it returns to include (but may be indicated). Nephritis if event if event does not improve with symptomatic treatment creatinine monitoring per protocol. Imited to): Renal treatment Systemic corticosteroids at a dose of 1-2 failure • Fatigue Renal treatment Systemic corticosteroids at a dose of 1-2 onsider • Increased equivalent may be indicated. When symptoms improve to Grade 1 or less, continued over at least 1 month. • Increased continued continued over at least 1 month. Consider prophylactic antibiotics for consider prophylactic antibiotics for continued over at least 1 month. • Swelling or creatinine creatinine creatinine creatinine continued boyer. Consider prophylactic antibiotics for consider prophylactic antibiotics for consider prophylactic antibiotics for consider prophylactic antibiotics for consider prophylactic antibiotics for consider prophylactic prophylactic antibiotics for consider prophylactic | Event(s) Grade I Consider • Provide symptomatic treatment. Symptoms may may include (but monitoring per protocol. Symptoms may include (but monitoring per protocol. Symptoms may include (but monitoring per protocol. Immited to): Immited to | Event(s) V4.03 Action/Supportive Care Guidelines Symptoms denal events Grade 1 Consider • Provide symptomatic treatment. Symptoms Nephritis if event • Discontinue • Provide symptomatic treatment. Image anto include (but not treatment. Nephritis if event • Discontinue • Provide symptomatic treatment not include to provide symptoms in the symptomatic treatment. • Imited to): Renal Grade 2 Consider • mg/kg/day of preduisone or equivalent may be indicated. When symptoms improve to Grade 1 or less, continued over at least 1 month. • Increased equivalent may be indicated. When symptoms improve to Grade 1 or less, continued over at least 1 month. • Increased equivalent may be indicated. When symptoms improve to Grade 1 or less, continued over at least 1 month. • Increased equivalent may be indicated. When symptoms improve to Grade 1 or less, continued over at least 1 month. • Increased equivalent may be indicated. When symptoms improve to Grade 1 or less, continued over at least 1 month. • Retailing Renal Grade 3- • Grade 4. • Grade 4. | Parent(s) Grade Consider Provide symptomatic treatment Monitor creatinine weekly, when it returns to include (but may withholding Provide symptomatic treatment Monitor creatinine weekly, when it returns to include (but may be buttern) Monitor creatinine weekly, when it returns to include (but may be indicated been not improve with symptomatic treatment Systemic corticosteroids at a dose of 1-2 Farigue Pressure Farigue Pressure Pre | Event(s) Grade of Grade Action/Supportive Care Guidelines Symptoms may be made that the consider of the consideration of the | Event(s) Grade 1 Grade 1 Consider • Provide symptomatic treatment. Symptoms may be upformed to the creatinine weekly; when it returns to include (but may be britis) autoimmune Provide symptomatic treatment. Provide symptomatic treatment. Symptoms may be creatinine weekly; when it returns to include (but not treatment does not improve with symptomatic treatment does not improve to treatment does not improve to treatment treatment. Provide symptomatic treatment may be indicated. Symptoms may be indicated. Immed to): | Provider Provide symptomatic treatment Nephritis Withholding Provide symptomatic treatment Nephritis MAMUNOTHERAPY Provide symptomatic treatment Manitor creatinine weekly; when it returns to include (but not not include (but n | Provide Symptomatic treatment Nephritis Withholding Withholding Provide symptomatic treatment Nephritis Withholding Provide symptomatic treatment Nephritis Withholding Provide symptomatic Passeline, resume routine Nithholding Provide symptomatic Passeline, resument Patient Passeline Passeline, resument Patient Passeline Pa | kenal Grade 1 Consider Provide symptomatic treatment Symptoms Nephritis Withholding - Provide symptomatic treatment - Provide symptomatic treatment Imited (but may may be made to the provide symptomatic treatment of the symptomatic treatment of the symptomatic treatment of the symptomatic treatment of the symptomatic treatment of the symptomatic or treatment of the symptomatic treatment of the symptomatic or treatment of the symptoms or treatment or tr | Provide Symptomatic treatment Symptoms | Grade Consider Provide symptomatic treatment Prestment continue weekly, when it returns to include (but autoimmune does not improve Prestment continue per protocol. Imited to): | Grade Consider Provide symptomatic treatment Consider Provide symptomatic treatment Consider Provide symptomatic autoimmune Consider Consider Provide symptomatic treatment Consider Cons | Crade Consider Provide symptomatic treatment Consider Provide symptomatic treatment Pragram Pra | Provide Symptomatic treatment Symptoms |

| Diagnosis | All attempts | should be made | to rule out other<br>causes such as | metastatic | disease,<br>infection, or | allergic<br>dermatitis. | | | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Action/Supportive Care Guidelines | Symptomatic treatment should be given such as topical glucocorticosteroids | (eg. octamentasoue 0.1% cream of hydrocortisone 1%) or urea-containing creams in combination with oral | antiprurities (e.g., diphenhydramine HCl<br>or<br>hydroxyzine HCl).<br>Treatment with oral steroids is at | investigator discretion for Grade 2. • events. | | | Consider dermatology consultation and biopsy for confirmation of diagnosis. Treatment with oral steroids is | recommended, starting with 1 mg/kg | predizione or equivalent once per day<br>or dexamethasone 4 mg four times | orally daily. When symptoms improve to Grade 1 or less, steroid taner | should be started and continued over no less than 4 weeks. | Dermatology consultation and consideration of biopsy and clinical | dermatology photograph. Initiate steroids at 1? mo/ke | prednisone or equivalent. When | improve to grade 1 or less, steroid taper<br>should be started and continued over | no less than 4 weeks. | | | Grade 3 drug-related thrombocytopenia >7 days or associated with bleeding | requires discontinuation. | Grade 4 drug-related thrombocytopenia > >7 days or associated with bleeding requires discontinuation | | |
| | No change in dose | | | | . 1000 | | Hold<br>IMMUNOTHERAPY. | | | | | Permanently | discontinue | IMMUNOTHERAPY. | | | No change in dose | No change in dose | No change in dose | *** | Hold<br>IMMUNOTHERAPY | < Grade 1. May | interval by 1 week. |
| v4.03<br>Grade | Grade 1–<br>2 | | | | | | Grade 3 | | | | | Grade 4 | | | | | ≤ Grade 1 | Grade 2 | Grade 3 | | Grade 4 | | |
| Event(s) | ents | Dermatitis | exfoliative<br>Erythema | multiforme<br>Stevens- | Johnson<br>syndrome<br>Toxic | epidermal<br>necrolysis | If considered to be | related, | ≥ Grade 3 or result | in dose modification | or discontinuation: | Pruritus | Rash | Rash<br>generalized | Rash<br>maculo- | papular<br>Vitiligo | Thrombocytopenia | • | | | | | |
| ( ) | Skin events | • | • | | • | • | If consic | immune related | ≥ Grade | in dose 1 | or discor | | ) | • | • | • | Thromk | | | | | | |

<sup>&</sup>lt;sup>a</sup> The signs and symptoms may be associated with any of the diagnoses in the associated "Event(s)" column.

<sup>b</sup> REMICADE (Infliximab) prescribing information

<sup>c</sup> If symptoms indicate possible new or worsening cardiac abnormalities, additional testing and/or a cardiology consultation should be considered.

**Table 3.0** OAR Dose Limits for 3 fraction SBRT

| Serial Organ | Volume | Volume Dose | Avoidance Endpoint |
|---|---|---|---|
| Spinal Cord | <0.03 cc | (Gy)<br>22.5 | Myelitis |
| | <1.2 cc | 13 | Myelitis |
| Ipsilateral Brachial Plexus | < 0.03 cc | 26 | Brachial Plexopathy |
| to the state of th | 8 | 22 | Brachial Plexopathy |
| Cauda Equina | <0.03 cc | 25.5 | Neuritis |
| | \$\$ | 21.9 | Neuritis |
| Sacral Plexus | <0.03 cc | 24 | Neuropathy |
| | 33 \$> | 22.5 | Neuropathy |
| Trachea and Ipsilateral<br>Bronchus* | <0.03 cc | 30 | Stenosis/Fistula |
| | <500 | 25.8 | Stenosis/Fistula |
| Esophagus* | <0.03 cc | 27 | Stenosis/Fistula |
| 1.7.1004.64 | <5cc | 17.7 | Stenosis/Fistula |
| Heart/Pericardium | <0.03cc | 30 | Pericarditis |
| The state of the s | <15 cc | 24 | Pericarditis |
| Great vessels* | <0.03cc | 45 | Aneurysm |
| | <10 cc | 39 | Aneurysm |
| Skin | <0.03cc | 33 | Ulceration |
| | <10cc | 31 | Ulceration |
| Stomach | <0.03cc | 30 | Ulceration/Fistula |
| | <10cc | 22.5 | Ulceration/Fistula |
| Duodenum* | <0.03cc | 24 | Ulceration |
| The second secon | | T | |

| | <10cc | 15 | Ulceration |
|---|---|---|---|
| Bowel* | <0.03 cc | 34.5 | Ulceration |
| | <20cc | 24 | Colitis/Fistula |
| Rectum* | <0.03 € | 49.5 | Ulceration |
| | <3.5 cc | 45 | Proctitis/Fistula |
| | < 20 cc | 27.5 | Proctitis/Fistula |
| Bladder | 0.03cc | 33 | Cystitis/Fistula |
| | <15 cc | 16.8 | Cystitis/Fistula |
| Ureter | <0.03 cc | 40 | Stenosis |
| Penile bulb | <3cc | 25 | Impotence |
| Femoral heads | <10 cc | 24 | Necrosis |
| Bile duct | < 0.03 cc | 36 | Stenosis |
| Renal hilum/vascular trunk | <15 cc | 19.5 | Malignant Hypertension |
| Rib | < 0.03 cc | 50 | Pain or Fracture |
| | <5 cc | 40 | Pain or Fracture |
| Parallel Organ | Volume | Volume Dose<br>(Gy) | Avoidance Endpoint |
| Lung (total) | <15% lung<br>volume | 20 | Pneumonitis/Lung Function |
| | < 37% lung<br>volume | 11 | Pneumonitis |
| | 1500 cc | 10.5 | Basic Lung Function |
| - Communication of the Communi | 1000 cc | 11.4 | Pneumonitis |
| Ipsilateral kidney | <130 cc | 12.3 | Nephritis |
| Total Kidney | <200cc | 15 | Basic Renal Function |
| Liver | <700 cc | 17.1 | Liver function |
| *NOTE: Avoid circumfarantial irradiation | TO THE PERSON NAMED IN COLUMN TWO IS NOT THE PERSON NAMED IN COLUMN TW | | |

<sup>\*</sup>NOTE: Avoid circumferential irradiation.

Table 4.0 OAR Dose Limits for 5 fraction SBRT

| Serial Organ | Volume | Volume Dose (Gy) | Avoidance |
|---|---|---|---|
| 7 | | | Endpoint |
| Spinal Cord | <0.03 cc | 28 | Myelitis |
| | <0.35 cc | 22 | Myelitis |
| | <1.2 cc | 15.6 | Myelitis |
| Ipsilateral Brachial Plexus | < 0.03 cc | 32 | Brachial<br>Plexopathy |
| | \$<br>8 | 30 | Brachial<br>Plexopathy |
| Cauda Equina | <0.03 cc | 32 | Neuritis |
| | % € | 30 | Neuritis |
| Sacral Plexus | <0.03 cc | 32 | Neuropathy |
| | 33 \$> | 30 | Neuropathy |
| Trachea and Ipsilateral Bronchus* | <0.03cc | 40 | Stenosis/Fistula |
| | 335> | 32 | Stenosis/Fistula |
| Esophagus* | <0.03cc | 35 | Stenosis/Fistula |
| | > € | 27.5 | Stenosis/Fistula |
| Heart/Pericardium | <0.03 cc | 38 | Pericarditis |
| The state of the s | <15 cc | 32 | Pericarditis |
| Great vessels* | <0.03 cc | 53 | Aneurysm |
| | <10 cc | 47 | Aneurysm |
| Skin | < 0.03cc | 38.5 | Ulceration |
| | <10cc | 36.5 | Ulceration |
| Stomach | > 0.5cc | 35 | Ulceration |
| | 205> | 26.5 | Ulceration |
| Duodenum* | < 0.5 cc | 30 | Ulceration |

| TOTAL PROPERTY OF THE PROPERTY | | | |
|---|---|---|---|
| | < 5 cc | 18.3 | Ulceration |
| Bowel* | < 0.03 cc | 40 | Ulceration |
| | <20 cc | 28.5 | Colitis/Fistula |
| Rectum* | <0.03 cc | 55 | Ulceration |
| | <3.5 cc | 50 | Proctitis/Fistula |
| | <20 cc | 32.5 | Proctitis/Fistula |
| Bladder | < 0.03 | 38 | Cystitis/Fistula |
| | <15 cc | 20 | Cystitis/Fistula |
| Ureter | < 0.03 cc | 45 | Stenosis |
| Penile Bulb | ~3 cc | 30 | Impotence |
| Femoral head | <10 cc | 30 | Necrosis |
| Bile Duct | <0.03 cc | 41 | Stenosis |
| Renal hilum/Vascular Trunk | <15 cc | 23 | Malignant<br>Hypertension |
| Rib | <0.03 cc | 57 | Pain or Fracture |
| | <5 cc | 45 | Pain or Fracture |
| Parallel Organ | Volume | Volume Dose (Gy) | Avoidance<br>Endpoint |
| Lung (total) | < 37% lung<br>volume | 13.5 | Pneumonitis |
| | < 1500 cc | 12.5 | Basic Lung<br>Function |
| , puntation | < 1000 cc | 13.5 | Pneumonitis |
| Total Kidney | < 200cc | 18 | Basic Renal<br>Function |
| Liver | <700 cc | 21 | Liver Function |
| THE RESERVE THE PROPERTY OF THE PARTY OF THE | | | |

\*NOTE: Avoid circumferential irradiation.

## APPENDIX III: STUDY PARAMETERS AND ASSESSMENTS

Table 5.0: Pre-treatment assessments

| Assessment | Time Points |
|---|---|
| | ≤30 days prior to registration |
| Evaluation by a radiation oncologist | X |
| Evaluation by a medical oncologist | X |
| History/physical examination | X |
| Performance Status<br>(ECOG) | X |
| CBC w/ diff & ANC,<br>platelets, ALT, AST | ≤ 30 days prior to registration <u>.</u> |
| Serum/urine<br>pregnancy test (if<br>applicable) | $\leq 14$ days prior to registration |
| CT Scans of the chest/abdomen/ pelvis with radionuclide bone scan OR whole body PET/CT | × |
| Histological<br>confirmation from at<br>least one metastasis | X |
| MRI of the vertebral<br>column | If vertebral column metastases identified on staging and will be treated |

Table 6.0: Post-Treatment Assessments

## ASSESSMENTS IN FOLLOW-UP

| Assessment | Time Points | ots |
|---|---|---|
| | 30 days after completion of SBRT | Every 3 months after<br>completion of SBRT for a<br>total of 2 years |
| Physical examination | X | X |
| Evaluation by a radiation<br>oncologist | X | × |
| Performance status | X | X |
| ALT, AST, Total and Direct<br>Bilirubin | X r. r. ii.e managan | X<br>(If SBRT delivered to the liver)<br>Perform at 3 months then every |
| | (If SBRT delivered to the liver) | 6 months |
| Hgb | Recommended if clinical symptoms of anemia on physical exam post-treatment | |
| Diagnostic Imaging | | X Per protocol or if clinically warranted |
| Adverse event evaluation | X | X |

# LIST OF COMMON ABBREVIATIONS AND DEFINITIONS OF TERMS

ADL Activities of Daily Living

AE Adverse event

AESI Adverse event of special interest

ALP Alkaline phosphatase

ALT Alanine aminotransferase

ANA Antinuclear antibody

ANC Absolute neutrophil count

aPTT Activated partial thromboplastin time

ARGUS Pharmacovigilance and clinical safety software system

AST Aspartate aminotransferase

AUC Area under the concentration-time curve

BAL Bronchoalveolar lavage

BC Breast cancer

BUN Blood urea nitrogen

CPA Cyclophosphamide

CR Complete response

CRF; eCRF Case report form (electronic or paper); electronic case report form

CRO Contract research organization

CRP C-reactive protein

CT Computed tomography

CTLA-4 Cytotoxic T-lymphocyte antigen 4

CTV Clinical target volume

(NCI-) CTCAE (National Cancer Institute) Common Terminology Criteria for Adverse Events

DLT Dose-limiting toxicity

Dmax Maximum radiation dose

EC Ethics committee

ECG Electrocardiogram

EDC Electronic data capture

FDG-PET 18F-fluorodeoxyglucose positron emission tomography

FFPE Formalin-fixed, paraffin-embedded

FNA Fine-needle aspirate

fx Fraction(s)

GCP Good clinical practice

GBM Glioblastoma multiforme

GM-CSF Granulocyte-macrophage colony-stimulating factor

GTV Gross target volume

H&N Head and neck

HPV human papillomavirus

HLA Human leukocyte antigen

ICF Informed consent form

ICH International Conference on Harmonisation

IHC Immunohistochemistry

INR International Normalized Ratio

irRC Immune-related response criteria

IRB Institutional Review Board

irAE Immune-related adverse event

ITV. Internal target volume

IUD Intrauterine device

IV Intravenous

LC Local control

LD Longest diameter

LE Local enlargement

LDH Lactate dehydrogenase

LDL Low-density lipoprotein

LLOQ Lower limit of quantification

mAb Monoclonal antibody

Max Vol Maximum (tissue) volume

MedDRA Medical Dictionary for Regulatory Activities

monoRX Monotherapy

MRI Magnetic resonance imaging

MTD Maximum tolerated dose

NCI-CTCAE National Cancer Institute-Common Terminology Criteria for Adverse Events

NOAEL No-observed-adverse-effect level

NSCLC Non-small-cell lung cancer

PBMC Peripheral blood mononucleated cell

PD-1 Programmed death-1 (receptor)

PD-L1, PD-L2 Programmed death ligand 1, programmed death ligand 2

PET Positron-emission tomography

PK Pharmacokinetic

PR Partial response

PT Preferred term

PTV Planning target volume

RBC Red blood cell

RCC Renal cell cancer

RECIST Response Evaluation Criteria in Solid Tumors

Regeneron Regeneron Pharmaceuticals, Inc.

RF Rheumatoid factor

RILD Radiation-induced liver disease

RP2D Recommended phase 2 dose

SAE Serious adverse event

SAF Safety analysis set

SAP Statistical analysis plan

SAS Statistical Analysis Systems (software)

SABR Stereotactic Ablative Radiatiotherapy

SBRT Stereotactic Body Radiotherapy

SCHNC squamous-cell head and neck cancer

SOC System organ class

SSA Sjögren's syndrome A antigen

SSB Sjögren's syndrome B antigen

t1/2 Beta-phase terminal half life

TEAE Treatment-emergent adverse event

TSA a mouse mammary adenocarcinoma cell line

TSH Thyroid-stimulating hormone

WBC White blood cell

XRT Radiotherapy

#### REFERENCES

- Mittal D, Gubin MM, Schreiber RD, et al.: New insights into cancer immunoediting and its three component phases--elimination, equilibrium and escape. Curr Opin Immunol 27:16-25,
- Schreiber RD, Old LJ, Smyth MJ: Cancer immunoediting: integrating immunity's roles in cancer suppression and promotion. Science 331:1565-1570, 2011 d
- Vesely MD, Kershaw MH, Schreiber RD, et al.: Natural innate and adaptive immunity to cancer. Annu Rev Immunol 29:235-271, 2011 ઌ
- Hanahan D, Weinberg RA: Hallmarks of cancer: the next generation. Cell 144:646-674, 2011 4.
- Zou W, Chen L: Inhibitory B7-family molecules in the tumour microenvironment. Nat Rev Immunol 8:467-477, 2008 Ś.
- Creelan BC: Update on immune checkpoint inhibitors in lung cancer. Cancer Control 21:80-89, 6
- Wei B, Wang L, Zhao X, et al.: The upregulation of programmed death 1 on peripheral blood T cells of glioma is correlated with disease progression. Tumour Biol 35:2923-2929, 2014 7
- Zandberg DP, Strome SE: The role of the PD-L1:PD-1 pathway in squamous cell carcinoma of the head and neck. Oral Oncol 50:627-632, 2014 ∞
- Francisco LM, Sage PT, Sharpe AH: The PD-1 pathway in tolerance and autoimmunity. Immunol Rev 236:219-242, 2010 6
- Topalian SL, Hodi FS, Brahmer JR, et al.: Safety, activity, and immune correlates of anti-PD-1 antibody in cancer. N Engl J Med 366:2443-2454, 2012 10.
- Lock M, Muinuddin A, Kocha WI, et al.: Abscopal Effects: Case Report and Emerging Opportunities. Cureus 7:e344, 2015 Ξ:
- Formenti SC, Demaria S: Combining radiotherapy and cancer immunotherapy: a paradigm shift. J Natl Cancer Inst 105:256-265, 2013 12.
- Tang C, Wang X, Soh H, et al.: Combining radiation and immunotherapy: a new systemic therapy for solid tumors? Cancer Immunol Res 2:831-838, 2014 13.
- immunogenic tumor cell death by ionizing irradiation implications for cancer therapies. 14. Frey B, Rubner Y, Wunderlich R, et al.: Induction of abscopal anti-tumor immunity and Curr Med Chem 19:1751-1764, 2012
- Bezu L, Gomes-de-Silva LC, Dewitte H, et al.: Combinatorial strategies for the induction of immunogenic cell death. Front Immunol 6:187, 2015 15.
- Kwilas AR, Donahue RN, Bernstein MB, et al.: In the field: exploiting the untapped potential of immunogenic modulation by radiation in combination with immunotherapy for the treatment of cancer. Front Oncol 2:104, 2012 16.
- Garnett CT, Palena C, Chakraborty M, et al.: Sublethal irradiation of human tumor cells modulates phenotype resulting in enhanced killing by cytotoxic T lymphocytes. Cancer Res 64:7985-17.
- McFarland HI, Puig M, Grajkowska LT, et al.: Regulatory T cells in gamma irradiation-induced immune suppression. PLoS One 7:e39092, 2012 18.
- induces an immune-mediated abscopal effect when combined with anti-CTLA-4 antibody. Dewan MZ, Galloway AE, Kawashima N, et al.: Fractionated but not single-dose radiotherapy Clin Cancer Res 15:5379-5388, 2009 19.
- Derer A, Deloch L, Rubner Y, et al.: Radio-Immunotherapy-Induced Immunogenic Cancer Cells as Basis for Induction of Systemic Anti-Tumor Immune Responses Pre-Clinical Evidence and Ongoing Clinical Applications. Front Immunol 6:505, 2015 20.
- 21. Lee Y, Auh SL, Wang Y, et al.: Therapeutic effects of ablative radiation on local tumor require CD8+ T cells. changing strategies for cancer treatment. Blood 114:589-595, 2009
- Pilones KA, Vanpouille-Box C, Demaria S: Combination of radiotherapy and immune checkpoint inhibitors. Semin Radiat Oncol 25:28-33, 2015 22.
- Kalbasi A, June CH, Haas N, et al.: Radiation and immunotherapy: a synergistic combination. J Clin Invest 123:2756-2763, 2013 23.
- Demaria S, Pilones KA, Vanpouille-Box C, et al.: The optimal partnership of radiation and immunotherapy: from preclinical studies to clinical translation. Radiat Res 182:170-181, 24.
- radiation-induced antitumor responses with immunotherapy. Radiat Res 182:126-138, 2014 Wattenberg MM, Fahim A, Ahmed MM, et al.: Unlocking the combination: potentiation of 25.
- definitive radiotherapy in patients with localized prostate cancer. Clin Cancer Res 11:3353-3362, 2005 Gulley JL, Arlen PM, Bastian A, et al.: Combining a recombinant cancer vaccine with standard 26.
- Hodge JW, Sharp HJ, Gameiro SR: Abscopal regression of antigen disparate tumors by antigen cascade after systemic tumor vaccination in combination with local tumor radiation. Cancer Biother Radiopharm 27:12-22, 2012 27.
- Anestakis D, Petanidis S, Kalyvas S, et al.: Mechanisms and applications of interleukins in cancer immunotherapy. Int J Mol Sci 16:1691-1710, 2015 28.
- Kachikwu EL, Iwamoto KS, Liao YP, et al.: Radiation enhances regulatory T cell representation. Int J Radiat Oncol Biol Phys 81:1128-1135, 2011 29.

- Wei S, Egenti MU, Teitz-Tennenbaum S, et al.: Effects of tumor irradiation on host T-regulatory cells and systemic immunity in the context of adoptive T-cell therapy in mice. J Immunother 36:124-132, 2013 30.
- McDermott DF, Atkins MB: PD-1 as a potential target in cancer therapy. Cancer Med 2:662-673, 2013
- Deng L, Liang H, Burnette B, et al.: Irradiation and anti-PD-L1 treatment synergistically promote antitumor immunity in mice. J Clin Invest 124:687-695, 2014 32.
- Sharabi AB, Nirschl CJ, Kochel CM, et al.: Stereotactic Radiation Therapy Augments Antigen-Specific PD-1-Mediated Antitumor Immune Responses via Cross-Presentation of Tumor Antigen. Cancer Immunol Res 3:345-355, 2015 33.
- Zeng J, See AP, Phallen J, et al.: Anti-PD-1 blockade and stereotactic radiation produce long-term survival in mice with intracranial gliomas. Int J Radiat Oncol Biol Phys 86:343-349, 2013 34.
- Park SS, Dong H, Liu X, et al.: PD-1 Restrains Radiotherapy-Induced Abscopal Effect. Cancer Immunol Res 3:610-619, 2015 35.
- Brahmer J, Reckamp KL, Baas P, et al.: Nivolumab versus Docetaxel in Advanced Squamous-Cell Non-Small-Cell Lung Cancer. N Engl J Med 373:123-135, 2015 36.
- Rusthoven KE, Hammerman SF, Kavanagh BD, et al.: Is there a role for consolidative stereotactic body radiation therapy following first-line systemic therapy for metastatic lung cancer? A patterns-of-failure analysis. Acta Oncol 48:578-583, 2009
- patients with one to five sites of metastatic disease. Clin Cancer Res 14:5255-5259, 2008 Salama JK, Chmura SJ, Mehta N, et al.: An initial report of a radiation dose-escalation trial in 38.
- Sheu T, Heymach JV, Swisher SG, et al.: Propensity score-matched analysis of comprehensive local therapy for oligometastatic non-small cell lung cancer that did not progress after front-line chemotherapy. Int J Radiat Oncol Biol Phys 90:850-857, 2014 39.
- therapy or observation for patients with oligometastatic non-small-cell lung cancer without Gomez DR, Blumenschein GR, Jr., Lee JJ, et al.: Local consolidative therapy versus maintenance progression after first-line systemic therapy: a multicentre, randomised, controlled, phase study. Lancet Oncol, 2016 40.
- Steven Chmura: Stereotactic Body Radiation Therapy in Treating Patients With Metastatic Breast Cancer, Non-small Cell Lung Cancer, or Prostate Cancer, in , 2016 41.

## STUDY ADDENDUM 1.

progression free survival, 6 month overall survival and response rate were significantly improved Additional immunotherapy agents have shown efficacy in the treatment of metastatic NSCLC in the first line setting. Pembrolizumab is a humanized monoclonal antibody against the PD-1 with and no sensitizing mutation of the epidermal growth factor receptor gene or translocation of the in the Pembrolizumab arm. Pembrolizumab has now redefined initial systemic therapy for PDanaplastic lymphoma kinase gene to receive either Pembrolizumab (at a fixed dose of 200 mg previously untreated advanced NSCLC with PD-L1 expression on at least 50% of tumor cells Since the development of this study, additional data regarding immunotherapy has emerged. antitumor activity in advanced NSCLC expressing PD-L1. The Keynote-024 trial compared every 3 weeks) or the investigator's choice of platinum-based chemotherapy (1). Median L1 expressing tumors in the metastatic setting.

We hereby propose that immunotherapy in this trial now include Nivolumab or Pembrolizumab as long as patients are eligible.

#### References

1. Reck M et al. N Engl J Med. 2016 Nov 10;375(19):1823-1833. Epub 2016 Oct 8.

## STUDY ADDENDUM 2.

immunotherapy landscape from randomized phase III trials. These changes affect our proposed utilization of stereotactic body radiation therapy (SBRT) and immunotherapy in 17-009 Since the last re-authorization of the study, there have been several changes in the

increase in overall survival in patients with stage III non-small cell carcinoma when Darvalumab pembrolizumab/alimta and carboplatin vs carboplatin/alimta alone (1). This survival benefit was Similarly, Key-407 showed an improved overall survival in patients with metastatic squamous higher with increasing PD-L1 expression but was maintained regardless of PD-L1 expression. alone (2) with PD-L1 expression ≥1%. Additionally, the PACIFIC trial showed an significant cell lung carcinoma with combination carboplatin/taxol/pembrolizumab vs carboplatin/taxol chemotherapy and immunotherapy. Keynote-189 showed an improved overall survival with First line systemic therapy for metastatic lung adenocarcinoma now includes combination was added following concurrent chemoradiation vs observation (3).

With these changes in the immunotherapy landscape, it is highly likely that patients with lung cancer will be increasingly exposed to immunotherapy agents earlier in the treatment course making them ineligible for our study since we currently exclude patients with prior immunotherapy treatments. Early data with sequential or combination SBRT suggest increased immunotherapy efficacy with similar rates or minimal changes in the toxicity profile of immunotherapy agents (4-5). Since our initial eligibility criteria was designed to limit excess patient toxicity and current available data suggests a combination/sequential regimen is safe, it is prudent that we revise our inclusion/exclusion criteria.

We hereby propose that patients with prior/ongoing immunotherapy treatment be eligible for participation in this study. The eligibility criterion has been modified as such to reflect this

#### References

- Ghandi L. et al. Pembrolizumab plus Chemotherapy in Metastatic Non-Small-Cell Lung Cancer. N Engl J Med May 2018; 378:2078-2092
- Lopes G. et al. Pembrolizumab (pembro) versus platinum-based chemotherapy (chemo) score (TPS)  $\geq$  1%: Open-label, phase 3 KEYNOTE-042 study. J Clin Oncol 36, 2018 as first-line therapy for advanced/metastatic NSCLC with a PD-L1 tumor proportion (suppl; abstr LBA4).
- AstraZeneca Press Release 05/2018: https://www.astrazeneca.com/media-centre/pressreleases/2018/imfinzi-significantly-improves-overall-survival-in-the-phase-iii-pacifictrial-for-unresectable-stage-iii-non-small-cell-lung-cancer-25052018.html

- radiotherapy (SBRT) versus pembrolizumab alone in patients with advanced non-small Theelen W. et al. Randomized phase II study of pembrolizumab after stereotactic body cell lung cancer: The PEMBRO-RT study. J Clin Oncol 36, 2018 (suppl; abstr 9023) 4.
- McArthur H. et al. A phase II, single arm study assessing the  $e\square$  cacy of pembrolizumab (Pembro) plusradiotherapy (RT) in metastatic triple negative breast cancer (mTNBC). J Clin Oncol 36, 2018 (suppl; abstr 9023) 5.

PCK-01

## CLINICAL STUDY PROTOCOL

Protocol Title: A PROSPECTIVE TRIAL OF IMMUNOTHERAPY AND STEREOTACTIC CANCER: SBRT SENSITIZATION OF THE PROGRAMMED DEATH-1 (PD-1) EFFECT BODY RADIOTHERAPY (SBRT) FOR THE TREATMENT OF METASTATIC LUNG

VERSION 6.0, 06/18/2018

Clinical Phase: Pilot/Phase II

response should translate to increased progression free survival and improved survival relative to Hypothesis: The addition of Stereotactic Body Radiation Therapy sequenced prior to PD-1/PD-L1 blockade leads to increased immunogenicity and immune system response. Increased PD-1 blockade monotherapy in metastatic lung cancer.

#### Principal Investigator

Olusola Obayomi-Davies MD

Department of Radiation Oncology

Crozer Keystone Health System/Philadelphia CyberKnife Center

2010 West Chester Pike, Havertown, PA 19083

## STUDY ADDENDUM 2.

immunotherapy landscape from randomized phase III trials. These changes affect our proposed utilization of stereotactic body radiation therapy (SBRT) and immunotherapy in 17-009. Since the last re-authorization of the study, there have been several changes in the

increase in overall survival in patients with stage III non-small cell carcinoma when Darvalumab pembrolizumab/alimta and carboplatin vs carboplatin/alimta alone (1). This survival benefit was Similarly, Key-407 showed an improved overall survival in patients with metastatic squamous higher with increasing PD-L1 expression but was maintained regardless of PD-L1 expression. alone (2) with PD-L1 expression ≥1%. Additionally, the PACIFIC trial showed an significant cell lung carcinoma with combination carboplatin/taxol/pembrolizumab vs carboplatin/taxol chemotherapy and immunotherapy. Keynote-189 showed an improved overall survival with First line systemic therapy for metastatic lung adenocarcinoma now includes combination was added following concurrent chemoradiation vs observation (3).

With these changes in the immunotherapy landscape, it is highly likely that patients with lung cancer will be increasingly exposed to immunotherapy agents earlier in the treatment course making them ineligible for our study since we currently exclude patients with prior immunotherapy treatments. Early data with sequential or combination SBRT suggest increased immunotherapy efficacy with similar rates or minimal changes in the toxicity profile of immunotherapy agents (4-5). Since our initial eligibility criteria was designed to limit excess patient toxicity and current available data suggests a combination/sequential regimen is safe, it is prudent that we revise our inclusion/exclusion criteria.

We hereby propose that patients with prior/ongoing immunotherapy treatment be eligible for participation in this study. The eligibility criterion has been modified as such to reflect this

# 1. REVISED PATIENT ELIGIBILITY AND CRITERIA

The target study population comprises patients with metastatic lung cancer who are eligible for an immunotherapy agent as monotherapy or combination therapy.

#### 1.1 Inclusion Criteria

- 1. Histologically or cytologically confirmed Stage IV NSCLC according to the 7th AJCC staging manual. Patients with recurrent disease after definitive treatment with surgery or concurrent chemoradiation are eligible.
- 2. Patients must be eligible for an immunotherapy agent as determined by treating medical oncologist. Patients who progress after drug therapy (3 months) for ALK, EGFR or ROS

immunotherapy are eligible if sites of progression are amenable to local therapy for control. mutation positive lung cancer are eligible. Patients who received prior combination immunotherapy or single agent monotherapy are eligible. Patients who progress on

- 3. At least 2 lesions that are safely amenable to SBRT/SABR.
- 4. ECOG ≥2.
- (RECIST) 1.1 criteria for response assessment or at least 1 lesion with FDG avidity and CT 5. At least 1 measurable lesion according to Response Evaluation Criteria in Solid Tumors correlate that can be monitored for PET-CT response by SUV Max increase or decrease.
- 6.  $\geq$ 18 years old.
- 7. Normal Hepatic and renal function.
- 8. Bone marrow reserve:
- a. ANC  $\ge 1.5 \times 10^9$ /L
- b. Hemoglobin >9.0 g/dL
- c. Platelet count  $\ge 75 \times 10^9 / L$
- 9. Ability to comply with follow-up visits and evaluations, treatment planning and studies and other study related procedures and visits.
- 10. Ability to sign informed consent.

#### 1.2 Exclusion Criteria

- 1. Patients with active CNS metastases. If metastases are treated and patients return to baseline and no steroids are required, patients are eligible.
- 2. Active, known or suspected auto-immune disease.
- 3. Patients with medical conditions that require systemic immunosuppression.
- 4. Patients with a history of interstitial lung disease.
- 5. Other active malignancy requiring intervention.
- 6. Prior lung radiation, with the only metastatic targets in the lungs.
- 7. Unresolved toxicity from prior chemotherapy or anti-cancer treatment.
- 8. Current or prior enrollment in clinical trial with an investigational drug within 4 weeks.

9. Pregnancy or positive pregnancy test.

#### References

- Ghandi L. et al. Pembrolizumab plus Chemotherapy in Metastatic Non-Small-Cell Lung Cancer. N Engl J Med May 2018; 378:2078-2092 i.
  - Lopes G. et al. Pembrolizumab (pembro) versus platinum-based chemotherapy (chemo) score (TPS)≥1%: Open-label, phase 3 KEYNOTE-042 study. J Clin Oncol 36, 2018 as first-line therapy for advanced/metastatic NSCLC with a PD-L1 tumor proportion (suppl; abstr LBA4). d
    - AstraZeneca Press Release 05/2018: https://www.astrazeneca.com/media-centre/pressreleases/2018/imfinzi-significantly-improves-overall-survival-in-the-phase-iii-pacifictrial-for-unresectable-stage-iii-non-small-cell-lung-cancer-25052018.html m
- radiotherapy (SBRT) versus pembrolizumab alone in patients with advanced non-small Theelen W. et al. Randomized phase II study of pembrolizumab after stereotactic body cell lung cancer: The PEMBRO-RT study. J Clin Oncol 36, 2018 (suppl; abstr 9023) 4
- McArthur H. et al. A phase II, single arm study assessing the e□cacy of pembrolizumab (Pembro) plusradiotherapy (RT) in metastatic triple negative breast cancer (mTNBC). J Clin Oncol 36, 2018 (suppl; abstr 9023) Š.

## CLINICAL STUDY PROTOCOL

Protocol Title: A PROSPECTIVE TRIAL OF IMMUNOTHERAPY AND STEREOTACTIC CANCER: SBRT SENSITIZATION OF THE PROGRAMMED DEATH-1 (PD-1) EFFECT BODY RADIOTHERAPY (SBRT) FOR THE TREATMENT OF METASTATIC LUNG

**VERSION 6.0, 06/18/2018** 

Clinical Phase: Pilot/Phase II

response should translate to increased progression free survival and improved survival relative to Hypothesis: The addition of Stereotactic Body Radiation Therapy sequenced prior to PD-1/PD-L1 blockade leads to increased immunogenicity and immune system response. Increased PD-1 blockade monotherapy in metastatic lung cancer.

#### Principal Investigator

Olusola Obayomi-Davies MD

Department of Radiation Oncology

Crozer Keystone Health System/Philadelphia CyberKnife Center

2010 West Chester Pike, Havertown, PA 19083

and must not be disclosed to anyone other than designees of Precision Radiation Oncology for conduct of the study, Confidential: This document contains confidential information that is the property of Precision Radiation Oncology clinical investigators and members of the Institutional Review Board.

## STUDY ADDENDUM 2.

immunotherapy landscape from randomized phase III trials. These changes affect our proposed utilization of stereotactic body radiation therapy (SBRT) and immunotherapy in 17-009. Since the last re-authorization of the study, there have been several changes in the

increase in overall survival in patients with stage III non-small cell carcinoma when Darvalumab pembrolizumab/alimta and carboplatin vs carboplatin/alimta alone (1). This survival benefit was Similarly, Key-407 showed an improved overall survival in patients with metastatic squamous higher with increasing PD-L1 expression but was maintained regardless of PD-L1 expression. alone (2) with PD-L1 expression ≥1%. Additionally, the PACIFIC trial showed an significant chemotherapy and immunotherapy. Keynote-189 showed an improved overall survival with cell lung carcinoma with combination carboplatin/taxol/pembrolizumab vs carboplatin/taxol First line systemic therapy for metastatic lung adenocarcinoma now includes combination was added following concurrent chemoradiation vs observation (3).

With these changes in the immunotherapy landscape, it is highly likely that patients with lung cancer will be increasingly exposed to immunotherapy agents earlier in the treatment course making them ineligible for our study since we currently exclude patients with prior immunotherapy treatments. Early data with sequential or combination SBRT suggest increased immunotherapy efficacy with similar rates or minimal changes in the toxicity profile of immunotherapy agents (4-5). Since our initial eligibility criteria was designed to limit excess patient toxicity and current available data suggests a combination/sequential regimen is safe, it is prudent that we revise our inclusion/exclusion criteria.

We hereby propose that patients with prior/ongoing immunotherapy treatment be eligible for participation in this study. The eligibility criterion has been modified as such to reflect this

# 1. REVISED PATIENT ELIGIBILITY AND CRITERIA

The target study population comprises patients with metastatic lung cancer who are eligible for an immunotherapy agent as monotherapy or combination therapy.

#### 1.1 Inclusion Criteria

- 1. Histologically or cytologically confirmed Stage IV NSCLC according to the 7th AJCC staging manual. Patients with recurrent disease after definitive treatment with surgery or concurrent chemoradiation are eligible.
- 2. Patients must be eligible for an immunotherapy agent as determined by treating medical oncologist. Patients who progress after drug therapy (3 months) for ALK, EGFR or ROS

PCK-01

immunotherapy are eligible if sites of progression are amenable to local therapy for control. mutation positive lung cancer are eligible. Patients who received prior combination immunotherapy or single agent monotherapy are eligible. Patients who progress on

- 3. At least 2 lesions that are safely amenable to SBRT/SABR.
- 4. ECOG ≥2.
- (RECIST) 1.1 criteria for response assessment or at least 1 lesion with FDG avidity and CT 5. At least 1 measurable lesion according to Response Evaluation Criteria in Solid Tumors correlate that can be monitored for PET-CT response by SUV Max increase or decrease.
- 6.  $\geq$ 18 years old.
- 7. Normal Hepatic and renal function.
- 8. Bone marrow reserve:
- a. ANC  $\ge 1.5 \times 10^9 / L$
- b. Hemoglobin ≥9.0 g/dL
- c. Platelet count  $\ge 75 \times 10^9/L$
- 9. Ability to comply with follow-up visits and evaluations, treatment planning and studies and other study related procedures and visits.
- 10. Ability to sign informed consent.

#### 1.2 Exclusion Criteria

- 1. Patients with active CNS metastases. If metastases are treated and patients return to baseline and no steroids are required, patients are eligible.
- 2. Active, known or suspected auto-immune disease.
- 3. Patients with medical conditions that require systemic immunosuppression.
- 4. Patients with a history of interstitial lung disease.
- 5. Other active malignancy requiring intervention.
- 6. Prior lung radiation, with the only metastatic targets in the lungs.
- 7. Unresolved toxicity from prior chemotherapy or anti-cancer treatment.
- 8. Current or prior enrollment in clinical trial with an investigational drug within 4 weeks.

9. Pregnancy or positive pregnancy test.

PCK-01

#### References

- Ghandi L. et al. Pembrolizumab plus Chemotherapy in Metastatic Non-Small-Cell Lung Cancer. N Engl J Med May 2018; 378:2078-2092
- Lopes G. et al. Pembrolizumab (pembro) versus platinum-based chemotherapy (chemo) score (TPS) ≥ 1%: Open-label, phase 3 KEYNOTE-042 study. J Clin Oncol 36, 2018 as first-line therapy for advanced/metastatic NSCLC with a PD-L1 tumor proportion (suppl; abstr LBA4). ri
- AstraZeneca Press Release 05/2018: https://www.astrazeneca.com/media-centre/pressreleases/2018/imfinzi-significantly-improves-overall-survival-in-the-phase-iii-pacifictrial-for-unresectable-stage-iii-non-small-cell-lung-cancer-25052018.html 'n
- radiotherapy (SBRT) versus pembrolizumab alone in patients with advanced non-small Theelen W. et al. Randomized phase II study of pembrolizumab after stereotactic body cell lung cancer: The PEMBRO-RT study. J Clin Oncol 36, 2018 (suppl; abstr 9023) 4;
- McArthur H. et al. A phase II, single arm study assessing the e□cacy of pembrolizumab (Pembro) plusradiotherapy (RT) in metastatic triple negative breast cancer (mTNBC). J Clin Oncol 36, 2018 (suppl; abstr 9023) 5